

# A 6-Week, Randomized Study to Evaluate the Potential of MC2-01 cream to Induce a Photoallergic Skin Reaction in Healthy Subjects, Using a Controlled Photopatch Test Design

Statistical Analysis Plan

Sponsor Protocol No. MC2-01-C10 TKL Study No. PB710518

08 April 2019

| Johan<br>Selmer | Digitally signed by Johan<br>Selmer<br>Date: 2019,04,09 12:52:31<br>+02'00' | |
|---|---|---|
| S | ignature | Date |
| S | ignature | Date |
| | Selmer | Selmer Selmer Date: 2019,04.09 12:52:31 |

# **TABLE OF CONTENTS**

| 1. STUDY PROTOCOL AND AMENDMENTS | 3 |
|---|---|
| 2. OBJECTIVES | 3 |
| 3. STUDY DESIGN | 3 |
| 4. DATA SETS | 4 |
| 5. HARDWARE AND SOFTWARE | 4 |
| 6. CODING | 5 |
| 7. STATISTICAL DATA REVIEW | 5 |
| B. HANDLING OF MISSING DATA | 5 |
| 9. DATABASE CLOSURE | 5 |
| 10. INTERIM AND SUBGROUP ANALYSES | 5 |
| 11. STATISTICAL EVALUATION | |
| 11.1 General Considerations for Data Analyses | |
| 11.2 Subject Populations for Analysis | |
| 11.2.1. Population I | |
| 11.2.2. Population II | |
| 11.2.3. Population III | |
| 11.3 Subject Disposition | |
| 11.4 Background and Demographic Characteristics | |
| 11.5 Study Products/Visit Compliance | |
| 11.6 Prior and Concomitant Therapy | |
| <ul><li>11.7 Dermal Response Evaluation</li><li>11.8 Safety Evaluation</li></ul> | |
| ~ <i></i> | |
| 11.9 Rationale for Selection of Sample Size | 10 |
| 12. CHANGES FROM THE PROTOCOL AND PLANNED ANALYSES | 10 |
| 13. HEADINGS | 10 |
| 14. ARCHIVING | 10 |
| 15. OUTLINE OF PROPOSED TABLES, FIGURES, AND LISTINGS | 11 |

# 1. STUDY PROTOCOL AND AMENDMENTS

This Statistical Analysis Plan is based on the Final Protocol dated 10 January 2019.

# 2. OBJECTIVES

The primary objective of this study will be to determine the photoallergic potential of MC2-01 cream when topical application to healthy skin is followed by light exposure. In addition, safety will be assessed by evaluation of any AEs reported during the study.

# 3. STUDY DESIGN

This will be a randomized, double-blind, single-center, controlled, within-subject comparison study of the investigational products (IPs), MC2-01 cream, MC2-01 vehicle, and an untreated irradiated control site in healthy volunteer subjects. A total of 8 application sites (2 cm x 2 cm each) will be marked on the subject's back and distributed so that 4 sites are on one side of the back for induction, and 4 sites are on the other side for challenge patches. The IPs will be applied in two sets. One set of patches on the back will be designated for irradiation after approximately 24 hours (± 4 hours) of study product application and the other set will remain non-irradiated. An additional site will be marked on the back during Challenge. The site will receive no treatment but will be irradiated at Challenge to serve as an untreated irradiated control.

A defined area (approximately 50 cm<sup>2</sup>) on the infrascapular region of each subject's back will be irradiated to determine the minimal erythemal dose (MED) of ultraviolet (UV) light.

During the 3-week Induction Phase of the study, 0.2 g of each study product will be applied to 2 sites twice each week (Monday and Thursday) for approximately 24 hours (± 4 hours) under semi-occlusive patch conditions (6 applications). After patch removal, all application sites will be evaluated, and one application site of each study product will be irradiated with 2 times the subject's MED using the full Xenon lamp spectrum. The sites will be evaluated by a trained evaluator. All sites will be reevaluated post irradiation, at approximately 48 hours later when irradiated on Tuesdays and at approximately 72 hours later when irradiated on Fridays except when irradiated on the last Friday of the Induction Phase or after the last make-up visit (if required), the sites will not be evaluated because these readings are not used for determination of photosensitization and any response will have subsided by Monday. These procedures will be performed each week for 3 weeks of the Induction Phase. Dermal reactions at the application sites will be evaluated using a visual scale that rates the degree of erythema, edema, and other signs of cutaneous irritation.

At the end of the Induction Phase, the subjects will enter a Rest Period of 10-17 days and then a Challenge Phase. One application/irradiation session may be missed during the Induction Phase. If a subject misses an irradiation session during the Induction Phase, an additional application/irradiation session will be scheduled the Monday of rest period (week 4).

At Challenge, each study product will be applied in an amount of 0.2 g to 2 naive sites once for approximately 24 hours (±4 hours) under semi-occlusive patches. After 24 hours (±4 hours) of product application, all sites will be evaluated, and one application site of each product and the additional untreated site will be irradiated. The sites will be examined for dermal reactions at approximately 24 hours (±4 hours), 48 hours (±4 hours), and 72 hours (±4 hours) post-irradiation. A Rechallenge should be performed if a cutaneous response observed during the Challenge Phase indicates possible photosensitization or at the discretion of the Investigator.

The safety endpoints for this study are irritation responses during the Induction Phase, positive responses at Challenge (ie, reactions indicative of a sensitization response) and AEs.

# 4. DATA SETS

The study database will be constructed and maintained by TKL Data Management in accordance with its standard operating procedures (SOPs) and the Sponsor's specifications. A data management plan (DMP), including database/screen design specifications, CRF review guidelines, coding instructions, and edit check specifications will be submitted to the Sponsor for review prior to data entry. When the database has been declared to be complete and accurate as per the DMP, the database will be locked (i.e., the database software will not allow any further additions to, removals from, or other edits of the database). All changes to the database after that time must be authorized by the Sponsor in writing and a database unlock form and then the re-lock form will be signed by both TKL and Sponsor. Study Data Tabulation Model (SDTM) datasets will be constructed from the raw data sets. Analysis datasets (ADaM) that are necessary for table analyses will be generated from SDTM.

The study SDTM and ADaM datasets will be taken as input to validated SAS programs which generate the report-ready tables and listings. Each output display will show the names of the data sets and SAS program used to produce it. Upon completion of the study report, the data sets will be provided to the sponsor as SAS XPT transport files. Data sets will be CDISC compliant. A CDISC compliant define.xml and annotated CRF for SDTM datasets will also be provided to the sponsor.

# 5. HARDWARE AND SOFTWARE

Statistical analysis will be performed following TKL SOP 03-02-04 Preparation of Tables and Listings for Statistical Reporting. All statistical analysis will be performed using SAS Version 9.2 or higher with program code prepared specifically for the project by qualified TKL statisticians and SAS programmers.

The SAS programs will generate rich-text-formatted (RTF) output with the "RTF" extension using the SAS Output Delivery System (ODS). The summary tables and listings will be formatted using the Courier New 9-point font. The RTF output is included in report documents prepared with Microsoft Word and converted to PDF format without typographical change.

# 6. CODING

The Medical Dictionary for Regulatory Activities (MedDRA, Version 22.0 2019) coding dictionary will be used for the assignment of system organ class and preferred terms to AEs. The WHO Drug Dictionary Enhanced (WHO DDE Version B 1Q19) will be used for assignment of preferred terms and drug classifications (i.e., Anatomic-Therapeutic-Chemical [ATC] subgroups) to concomitant medications, as described in the Data Management Plan (DMP).

# 7. STATISTICAL DATA REVIEW

Data verification activities to be performed prior to delivery of the SAS datasets to the project statistician are described in the approved DMP. After completion of the data verification activities, the SAS datasets will be delivered to the project statistician along with documentation of any unresolved queries and data conventions applied that are not fully explained in the data or the DMP. After delivery of the SAS datasets and prior to unblinding of the study data, the project statistician will perform completeness and self-consistency checks of the study data. Queries will be issued to the Data Manager and resolved before closure of the database.

# 8. HANDLING OF MISSING DATA

Missing values will not be imputed.

# 9. DATABASE CLOSURE

After completion of all data review procedures, validation of the project database, and approval of the final database in writing by the Sponsor, the database will be closed ("locked"). After the closure of the clinical database and authorization to unblind the study, the treatment codes will be merged to the analysis data sets. Any changes to data, coding, populations, or analysis plan after database closure must be approved by the Sponsor, in writing, and TKL management, and documented in the study archive with a detailed explanation of changes and reasons for changes.

# 10.INTERIM AND SUBGROUP ANALYSES

No interim or subgroup analyses are planned.

# 11.STATISTICAL EVALUATION

# 11.1 General Considerations for Data Analyses

The focus of the statistical analysis will be the comparison with controls of the photoallergic response to the investigational product. The parameter for photoallergy will be the mean numerical

equivalent score. The diagnosis of a reaction indicative of photosensitivity will be made by the Principal Investigator according to working criteria described in detail in the study protocol. Photosensitivity is not to be determined by statistical methods. However, a supportive statistical analysis of numerical photoirritation scores during the Induction Phase will be performed.

All statistical processing will be performed using the SAS® system (version 9.2).

# 11.2 Subject Populations for Analysis

Three analysis populations will be defined. All subjects who receive treatment will be evaluable for AEs (Population III). The evaluation of photosensitization will be based on all subjects who complete the challenge phase of the study (Population I). The analysis of local tolerability will be based off all subjects who complete the induction phase of the study (Population II).

# 11.2.1. Population I

Photosensitization potential for each test product site will be assessed only among subjects completing the Induction and Challenge Phases for that product. To be considered a complete case for a particular test product, a subject must have 6 applications/irradiation and no less than 11 **subsequent** readings during Induction, 10-17 days rest, and 1 application and at 3 post-irradiation evaluations during Challenge for that product. However, those subjects who demonstrate photosensitization, even though they have not completed all visits, will also be included in this population and will be evaluated. If subject's patch sites were discontinued because they were considered by the Investigator to be pre-photosensitized during Induction, this subject will not be included in this population for that test product.

# 11.2.2. Population II

Photoirritation potential for each test product will be assessed only among subjects completing the Induction Phase. To be considered a complete case for each test product, a subject must have 6 applications/irradiation as scheduled in the Induction Phase and no less than 11 **subsequent** readings as scheduled during the Induction Phase for that product.

# 11.2.3. Population III

This population will include all subjects who received the study products. This will also be the population used for adverse events analyses.

# 11.3 Subject Disposition

The number of subjects screened, randomized, completing the Induction phase, completing the Challenge phase, included in the analysis of photosensitization (Population I), included in the

analysis of photoirritation (Population II), included in the analysis of adverse events (Population III) and discontinued (by reason for discontinuation) will be summarized using descriptive statistics.

# 11.4 Background and Demographic Characteristics

Descriptive statistics will be used to summarize demographic characteristics (i.e., age, gender, ethnicity, and race) and background characteristics (i.e. Fitzpatrick skin type and MED) for the randomized subject population. Past/coexistent medical history information for all randomized subjects will be presented in a by-subject listing. Urine pregnancy test results will be presented in a by-subject listing.

# 11.5 Study Products/Visit Compliance

Descriptive statistics will be used to summarize study product compliance for the randomized subject population.

# 11.6 Prior and Concomitant Therapy

Prior and concomitant medication information for all randomized subjects will be presented in a bysubject listing.

# 11.7 Dermal Response Evaluation

The following scoring grades and notations will be used for the evaluation of dermal response at each application and control site throughout the Induction and Challenge Phases of the study. Tape related irritation will not be graded as an irritant response at the patch site.

# **Grading of Responses**

| Response | Symbol | Numerical Equivalent<br>Score |
|---|---|---|
| Erythema | | |
| No reaction | - | 0 |
| Mild, but definite erythema | + | 1.0 |
| Moderate erythema | ++ | 2.0 |
| Marked/severe erythema | +++ | 3.0 |
| Edema | | |
| No reaction<br>Mild, but definite edema | 0 | 0<br>1.0 |
| Definite edema with erosion/vesiculation | ** | 2.0 |

# **Response Notations**

| Response/Comment | Notation |
|---|---|
| Hyperpigmentation | Hr |
| Hypopigmentation | Но |
| Vesiculation | V |
| Papular response | p |
| Papulovesicular response | pv |
| Damage to epidermis: oozing, crusting and/or superficial erosions | D |
| Itching | I |
| Spreading of reaction beyond patch study site (i.e., reaction where material | S |
| did not contact skin) | |
| Follicular irritation with or without pustule formation (folliculitis) | f |
| Subject absent | X |
| Patch dislodged | PD |
| Not patched | NP |
| No reaction | 0 |

Note: The numerical score for edema is to be added to the numerical score for erythema. The literal notations in the second part of the table are not associated with additional numerical value.

All assigned scores during the study will be summarized using frequency counts by treatment at each time point. Erythema and edema scores will be summarized separately. All pairwise comparisons will be performed on the mean of the Induction Phase response scores using Fisher's least significant differences in the analysis of variance (ANOVA) with effects of subjects and treatment. The response score for each subject will be calculated by summing the erythema and edema score and then the mean of the response scores at each reading during the Induction Phase will be calculated for the subject. Pairwise differences will be tested only if the null hypothesis of a common mean score for all products is rejected at the 5% level.

In case of gross violations of the model assumptions (normality, homoscedasticity), non-parametric analysis will be performed. All assigned scores during Induction for each product will be ranked within subject and compared pairwise using Wilcoxon signed-rank test. Pairs to be compared include each test sample irradiated versus non-irradiated and all pairwise comparisons on each side.

# 11.8 Safety Evaluation

# **Assessment of Photosensitization Response**

The determination of dermal photosensitization potential will be based on specific scoring criteria derived from observations in the Challenge Phase of the study and confirmed in the Rechallenge Phase, if necessary. Criteria specified in the study protocol may cause the continuation of a subject into the Rechallenge Phase of the study. The diagnosis of a photosensitization response will be made by the Investigator based on review of the observed skin responses after Challenge. Photosensitivity will not be determined by statistical methods. All assigned scores during induction and challenge will be summarized by frequency counts by time point and treatment. The incidence of photosensitization reactions will be summarized by frequency counts for each treatment.

# **Local Tolerability Assessments**

The mean numerical equivalent score by subject and treatment, including all scores assigned during induction, will be analyzed in the analysis of variance (ANOVA) with factors subject and treatment. Selected pairwise comparisons will be performed in the context of the ANOVA. Pairs to be compared are: each test sample irradiated versus non-irradiated (MC2-01 cream irradiated versus non-irradiated; vehicle irradiated versus non-irradiated, and untreated control irradiated versus non-irradiated) and all pairwise comparisons on each side (MC2-01 cream versus vehicle; MC2-01 cream versus untreated control; and vehicle versus untreated control; all on both the irradiated and non-irradiated sides).

## **Adverse Events**

Adverse events will be summarized as an overall incidence of at least one event, incidence within body systems only, and incidence by body system and preferred term. Each subject will contribute only once (e.g., the first occurrence) to each of the rates, regardless of the number of occurrences (events) the subject experiences. Treatment-emergent AEs will be summarized and tabulated by the system organ class and preferred term, by severity (mild, moderate, severe) and by relationship to study product (none, possible, probable, or definite). Treatment-emergent will be defined as any AE with an onset date on or after the first study product administration date. Any event with a missing onset date will be included as a treatment-emergent AE. Deaths and SAEs will be listed by subject.

# 11.9 Rationale for Selection of Sample Size

The sample size of 50 evaluable subjects conforms to industry and regulatory standards for determination of irritation when topical application to skin is followed by light exposure.

# 12.CHANGES FROM THE PROTOCOL AND PLANNED ANALYSES

There are no changes from the planned analyses in the protocol.

# 13.HEADINGS

Each page of the analysis will show the Sponsor's name and study number. Report tables will be embedded in the MS Word report document from SAS program output without change. The footer of each table will show the name of the SAS program module which generated it, the names of all data sets providing input data in the program and the date and time the table was generated.

# 14.ARCHIVING

After finalization of the analysis, the following will be archived at TKL Research, Inc. and/or with the Sponsor:

- Randomization list
- Statistical Analysis Plan
- Data Management Plan
- Annotated CRF
- All SAS code used in the project for statistical analysis
- Final delivered tables and listings as included in the clinical study report
- Final SAS datasets, with full audit trail from initial data entry through final accepted version
- SDTM and ADaM data sets
- Define.xml
- Study data and analysis data reviewer guides for any unavoidable CDISC-checker errors or warnings
- Relevant Correspondence

# 15.OUTLINE OF PROPOSED TABLES, FIGURES, AND LISTINGS

# **Summary Tables**

| Table | |
|---|---|
| Number | Title |
| 14.1.1 | Summary of Subject Enrollment and Disposition |
| 14.1.2 | Summary of Subject Demographics and Baseline Characteristics |
| 14.1.3 | Summary of Study Product and Visit Compliance |
| 14.2.1.1 | Summary of Dermal Responses by Response Scores and Notations during Induction |
| 14.2.1.2 | Summary of Dermal Responses by Response Scores during Induction |
| 14.2.1.3 | Summary of Dermal Responses by Response Scores and Notations during Challenge |
| 14.2.1.4 | Summary of Dermal Responses by Response Scores during Challenge |
| 14.3.1.1 | Overall Summary of Adverse Events |
| 14.3.1.2* | Summary of Treatment-Emergent Adverse Events by Maximum Severity |
| 14.3.1.3* | Summary of Treatment-Emergent Adverse Events by Maximum Relationship |

<sup>\*</sup>Tables 14.3.1.2 and 14.3.1.3 will only be included if there are a sufficient number of Treatment-Emergent AEs for multiple classified AE tables.

# **Data Listings**

| Listing | |
|----------|------------------------------------------------------------|
| Number | Title |
| 16.1.7 | Subject Randomization |
| 16.2.1 | Subject Disposition and Population Inclusion |
| 16.2.2 | Protocol Deviations |
| 16.2.4.1 | Subject Demographics and Baseline Characteristics |
| 16.2.4.2 | Medical History |
| 16.2.4.3 | Prior and Concomitant Medications |
| 16.2.5 | MED Determination |
| 16.2.6.1 | Assessment of Dermal Responses during Induction |
| 16.2.6.2 | Assessment of Residual Dermal Responses at Relocated Sites |
| 16.2.6.3 | Assessment of Dermal Responses during Challenge |
| 16.2.7.1 | Adverse Events |
| 16.2.7.2 | Serious Adverse Events and Deaths |
| 16.2.8 | Urine Pregnancy Test Results |
| 16.2.9 | Comments |

MC2 Therapeutics
Page X of Y
Protocol No. MC2-01-C10

Table 14.1.1: Summary of Subject Enrollment and Disposition

| Number of Subjects Screened | XX |
|---|---|
| Screen Failures, n (%) [1] | XX (XX.X) |
| Reason Not Randomized, n (%) | |
| Inclusion X: XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XX (XX.X) |
| Exclusion X: XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XX (XX.X) |
| Other | XX (XX.X) |
| Etc. | |
| Number of Subjects Randomized | XX |
| Number of Subjects Completing Induction, n (%) | XX(XX.X) |
| Number of Subjects Completing Challenge, n (%) | XX (XX.X) |
| Subjects Included in Analysis of Photosensitization (Population I), n (%) | XXX (XX.X) |
| Subjects Included in Analysis of Photoirritation (Population II), n (%) | XXX (XX.X) |
| Subjects Included in Analysis of Adverse Events (Population III), n (%) | XXX (XX.X) |
| Number of Subjects Discontinued, n (%) | XX (XX.X) |
| Reason for Discontinuation, n (%) | · / |
| Protocol Violation | X (XX.X) |
| Withdrawal of informed consent | X(XX.X) |
| Etc. | |

Note: Percentages are relative to the number of randomized subjects except where otherwise specified.

[1] Percentage is relative to total number screened.

MC2 Therapeutics
Page X of Y

Table 14.1.2: Summary of Subject Demographics and Baseline Characteristics All Randomized Subjects

| A go (voors) | Moon (SD) | VV VV (V VV) |
|---|---|---|
| Age (years) | Mean (SD) | XX.XX (X.XX) |
| | Median | XX.X |
| | Minimum, Maximum | XX.X, XX.X |
| Gender, n (%) | Male | XX (XX.X) |
| | Female | XX (XX.X) |
| Race, n (%) | White | XX (XX.X) |
| (1.1) | Black or African American | XX (XX.X) |
| | Asian | XX (XX.X) |
| | American Indian or Alaskan Native | XX (XX.X) |
| | Native Hawaiian or Pacific Islander | XX (XX.X) |
| | Multiple: XXXX and XXXX | XX (XX.X) |
| Ethnicity, n (%) | Hispanic or Latino | XX (XX.X) |
| | Non-Hispanic or Latino | XX (XX.X) |
| Fitzpatrick Skin Type, n (%) [1] | I | XX (XX.X) |
| | II | XX (XX.X) |
| | III | XX (XX.X) |
| MED | Mean (SD) | X.XX (X.XX) |
| | Minimum, Maximum | X.XX, X.XX |

<sup>[1]</sup> I = Always burns easily, never tans; II = Always burns easily, tans minimally; III = Burns moderately, tans gradually

MC2 Therapeutics Protocol No. MC2-01-C10 Page X of Y

Table 14.1.3: Summary of Study Product and Visit Compliance All Randomized Subjects

| | Number of Subjects Applied with Study Product or Evaluated, n(%) | | |
|---|---|---|---|
| Number of Subjects Attending, n(%) | MC2-01 cream | MC2-01 vehicle | Untreated |
| Screening/Day 1 | xx (XX.XX) | xx (XX.XX) | xx (XX.XX |
| Induction Week 1/Study Day 1 Application | xx (XX.XX) | xx (XX.XX) | xx (XX.XX |
| Induction Week 1/Study Day 2 Evaluation | xx (XX.XX) | xx (XX.XX) | xx (XX.XX |
| Induction Week 1/Study Day 4 Evaluation/Application | xx (XX.XX) | xx (XX.XX) | xx (XX.XX |
| Induction Week 1/Study Day 5 Evaluation | xx (XX.XX) | xx (XX.XX) | xx (XX.XX |
| Induction Week 2/Study Day 8 Evaluation/Application | xx (XX.XX) | xx (XX.XX) | xx (XX.XX |
| Induction Week 2/Study Day 9 Evaluation | xx (XX.XX) | xx (XX.XX) | xx (XX.XX |
| Induction Week 2/Study Day 11 Evaluation/Application | xx (XX.XX) | xx (XX.XX) | xx (XX.XX |
| Induction Week 2/Study Day 12 Evaluation | xx (XX.XX) | xx (XX.XX) | xx (XX.XX |
| Induction Week 3/Study Day 15 Evaluation/Application | xx (XX.XX) | xx (XX.XX) | xx (XX.XX |
| Induction Week 3/Study Day 16 Evaluation | xx (XX.XX) | xx (XX.XX) | xx (XX.XX |
| Induction Week 3/Study Day 18 Evaluation/Application | xx (XX.XX) | xx (XX.XX) | xx (XX.XX |
| Induction Week 3/Study Day 19 Evaluation | xx (XX.XX) | xx (XX.XX) | xx (XX.XX |
| Challenge Week 6/Patch Application | xx (XX.XX) | xx (XX.XX) | xx (XX.XX |
| Challenge Week 6/Evaluation and Irradiation | xx (XX.XX) | xx (XX.XX) | xx (XX.XX |
| Challenge Week 6/24 Hour Post-Irradiation Evaluation | xx (XX.XX) | xx (XX.XX) | xx (XX.XX |
| Challenge Week 6/48 Hour Post-Irradiation Evaluation | xx (XX.XX) | xx (XX.XX) | xx (XX.XX |
| Challenge Week 6/72 Hour Post-Irradiation Evaluation/End of Study | xx (XX.XX) | xx (XX.XX) | xx (XX.XX |

Page X of Y

#### Statistical Analysis Plan

MC2 Therapeutics

Table 14.2.1.1: Summary of Dermal Responses by Response Scores and Notations During Induction Population II

| | MC2- | 01 cream | MC2- | 01 vehicle | Untreated |
|---|---|---|---|---|---|
| Response | Irradiated | Non-Irradiated | Irradiated | Non-Irradiated | Irradiated |
| Reading 1, n (%) | | | | | |
| Response Score (Sum of | | | | | |
| Erythema and Edema) | | | | | |
| 0 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 1 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx(xx.x) |
| 1 Hr | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 2 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| etc. | xx (xx.x) | xx(xx.x) | xx (xx.x) | xx(xx.x) | xx (xx.x) |
| [Reading 2, n (%)] to | | | | | |
| [Reading 11, n (%)] | | | | | |
| Response Score | | | | | |
| 0 | xx(xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx(xx.x) |
| etc | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |

#### **Scores:**

Erythema: 0 = No reaction; 1 = Mild, but definite erythema; 2 = Moderate erythema; 3 = Marked/severe erythema;

Edema: 0 = No reaction; 1 = Mild, but definite edema; 2 = Definite edema with erosion/vesiculation

#### **Notations**:

Hr = hyperpigmentation; Ho = hypopigmentation; V = vesiculation; p= Papular response; pv= Papulovesicular response; D= Damage to epidermis; oozing, crusting, and/or superficial erosions; I=Itching; S= Spreading of reaction beyond patch study site (i.e., reaction where material did not contact skin); f= Follicular irritation with or without pustule formation (folliculitis).; X=Subject absent; PD=Patch dislodged; NP = Not Patched; 0=No Reaction

MC2 Therapeutics
Page X of Y

Table 14.2.1.2: Summary of Dermal Responses by Response Scores During Induction (Part I)

Population II

| | MC2- | 01 cream | MC2- | 01 vehicle | Untreated |
|---|---|---|---|---|---|
| Response | Irradiated | Non-Irradiated | Irradiated | Non-Irradiated | Irradiated |
| Reading 1, n (%) | | | | | |
| Response Score (Sum of | | | | | |
| rythema and Edema) | | | | | |
| 0 | xx(xx.x) | xx (xx.x) | xx(xx.x) | xx (xx.x) | xx(xx.x) |
| 1 | xx(xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 2 | xx(xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx(xx.x) |
| 3 | xx(xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx(xx.x) |
| 4 | xx(xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx(xx.x) |
| etc. | xx (xx.x) | xx(xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| [Reading 2, n (%)] to | | | | | |
| [Reading 11, n (%)] | | | | | |
| desponse Score | | | | | |
| 0 | xx(xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| etc | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |

#### Scores:

Erythema: 0 = No reaction; 1 = Mild, but definite erythema; 2 = Moderate erythema; 3 = Marked/severe erythema;

Edema: 0 = No reaction; 1 = Mild, but definite edema; 2 = Definite edema with erosion/vesiculation

Note: P values are from an analysis of variance of the average numerical score over all Induction Phase readings, with effects of subject and treatment, using Fisher's least significant differences.

 $Generated \ on \ XX/XX/XX: XXXX \ by \ XXXXXXXX \ / \ Uses: \ XXXX, \ XXXX/ \ Reference \ listing: \ 16.X.X$ 


Table 14.2.1.2: Summary of Dermal Responses by Response Scores During Induction (Part II)

Population II

| | MC2-01 cream | | MC2-01 vehicle | | Untreated |
|---|---|---|---|---|---|
| | Irradiated | Non-Irradiated | Irradiated | Non-Irradiated | Irradiated |
| N | XX | XX | XX | XX | XX |
| Mean (SD) | x.xx(x.xx) | x.xx(x.xx) | x.xx(x.xx) | x.xx(x.xx) | x.xx(x.xx) |
| values | | | | | |
| vs MC2-01 cream Irr | | X.XXX | X.XXX | x.xxx | X.XXX |
| vs MC2-01 cream Non-Irr | | | X.XXX | X.XXX | X.XXX |
| vs MC2-01 vehicle Irr | | | | X.XXX | X.XXX |
| vs MC2-01 vehicle Non-Irr | | | | | X.XXX |
| vs Untreated Irr | | | | | |

Mean: The mean is the average of the response scores, where the response scores are calculated by summing the erythema and edema scores for each subject.

#### **Scores:**

Erythema: 0 = No reaction; 1 = Mild, but definite erythema; 2 = Moderate erythema; 3 = Marked/severe erythema; Edema: 0 = No reaction; 1 = Mild, but definite edema; 2 = Definite edema with erosion/vesiculation

Note: P values are from an analysis of variance of the average numerical score (sum of erythema and edema) over all Induction Phase readings, with effects of subject and treatment, using Fisher's least significant differences.


Table 14.2.1.3: Summary of Dermal Responses by Response Scores and Notations During Challenge Population I
(N=XXX)

| | MC2- | 01 cream | MC2-( | 1 vehicle | Untreated |
|---|---|---|---|---|---|
| Time Post-Irradiation | Irradiated | Non-Irradiated | Irradiated | Non-Irradiated | Irradiated |
| N Sensitized [1] | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 0 hours, n (%) | | | | | |
| -0 | xx (xx.x) | xx(xx.x) | xx (xx.x) | xx (xx.x) | xx(xx.x) |
| 24 hours, n (%)] to [72 hours, n (%)] | | | | | |
| Response Score | | | | | |
| (Sum of Erythema and Edema) | | | | | |
| 0 | xx(xx.x) | xx (xx.x) | xx(xx.x) | xx (xx.x) | xx (xx.x) |
| 1 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 1 Hr | xx(xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 2 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| etc. | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |

<sup>[1]</sup> Sensitization classification made by the PI based on Challenge and Re-challenge

## **Scores:**

Erythema: 0 = No reaction; 1 = Mild, but definite erythema; 2 = Moderate erythema; 3 = Marked/severe erythema;

Edema: 0 = No reaction; 1 = Mild, but definite edema; 2 = Definite edema with erosion/vesiculation

#### **Notations**:

Hr = hyperpigmentation; Ho = hypopigmentation; V = vesiculation; p= Papular response; pv= Papulovesicular response; D= Damage to epidermis; oozing, crusting, and/or superficial erosions; I=Itching; S= Spreading of reaction beyond patch study site (i.e., reaction where material did not contact skin); f= Follicular irritation with or without pustule formation (folliculitis).; X=Subject absent; PD=Patch dislodged; NP = Not Patched; 0=No Reaction


Table 14.2.1.4: Summary of Dermal Responses by Response Scores During Challenge Population I (N=XXX)

| | MC2- | 01 cream | MC2-0 | 01 vehicle | Untreated |
|---|---|---|---|---|---|
| Time Post-Irradiation | Irradiated | Non-Irradiated | Irradiated | Non-Irradiated | Irradiated |
| N Sensitized [1] | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 0 hours, n (%) | | | | | |
| -0 | xx (xx.x) | xx(xx.x) | xx (xx.x) | xx(xx.x) | xx (xx.x) |
| 24 hours, n (%)] to [72 hours, n<br>(%)] | | | | | |
| Response Score<br>(Sum of Erythema and Edema) | | | | | |
| 0 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 1 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 2 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 3 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 4 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| etc. | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |

<sup>[1]</sup> Sensitization classification made by the PI based on Challenge and Re-challenge

# **Scores:**

Erythema: 0 = No reaction; 1 = Mild, but definite erythema; 2 = Moderate erythema; 3 = Marked/severe erythema; Edema: 0 = No reaction; 1 = Mild, but definite edema; 2 = Definite edema with erosion/vesiculation

Page X of Y

# Statistical Analysis Plan

**MC2** Therapeutics


Table 14.3.1.1: Overall Summary of Adverse Events
Population III

| | (N = XX) |
|---|---|
| Subjects with Any AE, n (%) | XX (XX.X) |
| Number of AEs | XX |
| Subjects with Any Treatment-emergent AE (TEAE), n (%) | XX (XX.X) |
| Number of Treatment-emergent AEs | XX |
| Subjects with Any Treatment-related TEAE, n (%) [1] | XX (XX.X) |
| Number of Treatment-related TEAEs | XX |
| Subjects with Any Serious TEAE, n (%) | XX (XX.X) |
| Number of Serious TEAEs | XX |
| Subjects with Any Severe TEAE, n (%) | XX (XX.X) |
| Number of Severe TEAEs | XX |
| Subjects with Any Moderate TEAE, n (%) | XX(XX.X) |
| Number of Moderate TEAEs | XX |
| Subjects with Any Mild TEAE, n (%) | XX(XX.X) |
| Number of Mild TEAEs | XX |
| Subjects with Any TEAE Leading to Discontinuation of Study Medication, n (%) | XX (XX.X) |
| Number of TEAEs Leading to Discontinuation of Study Medication | XX |

<sup>[1]</sup> Treatment-related AEs include definitely related, probably related and possibly related.


# Table 14.3.1.2: Summary of Treatment-Emergent Adverse Events By Severity Population III

# All (n=x)

| Severity | No. Events | No. Subjects (%) |
|----------|------------|------------------|
| Mild | XX | xx (xx.x) |
| Moderate | xx | xx (xx.x) |
| Severe | XX | xx (xx.x) |

<sup>&</sup>lt;Programming note: sort AE tables by number of subjects.>


xx (xx.x)

All (n=x)

XX

# Table 14.3.1.3: Summary of Treatment-Emergent Adverse Events By Relationship Population III

| Relationship | No. Events | No. Subjects (%) |
|--------------------|------------|------------------|
| Definitely Related | xx | xx (xx.x) |
| Probably Related | xx | xx (xx.x) |
| Possibly Related | XX | xx (xx.x) |

 $Generated \ on \ XX/XX/XX:XXXX \ by \ XXXXXXX \ / \ Uses: \ XXXX, \ XXXX/ \ Reference \ listing: 16.X.X$ 

Not Related

<sup>&</sup>lt;Programming note: sort AE tables by number of subjects.>

MC2 Therapeutics


Listing 16.1.7: Subject Randomization All Randomized Subjects

| | Informed | Met all<br>Inclusion/Exclusion | | | Randomization [1] | |
|---|---|---|---|---|---|---|
| Subject Number | Consent Date | Criteria? | Randomization Date | Randomization Number | Site 1 | Site 2 |
| XX | XXXX-XX-XX | Yes | XXXX-XX-XX | XX | Α | В |
| XX | XXXX-XX-XX | Yes | XXXX-XX-XX | XX | В | A |
| XX | XXXX-XX-XX | Yes | XXXX-XX-XX | XX | A | В |
| XX | XXXX-XX-XX | Yes | XXXX-XX-XX | XX | В | A |
| XX | XXXX-XX-XX | Yes | XXXX-XX-XX | XX | В | A |

[1] A = MC2-01 cream; B = MC2-01 vehicle

Generated on XX/XX/XX:XXXX by XXXXXXX / Uses: XXXX, XXXX

Page X of Y


# Listing 16.2.1: Subject Disposition and Population Inclusion All Randomized Subjects

| | Date (Day [1]) of | | | | | | An | Analysis Population | |
|---|---|---|---|---|---|---|---|---|---|
| Subject<br>Number | Screening | Day 1 | Last Visit | Last Contact | End of Study Status | Number<br>of Days<br>in Study<br>[2] | Population I –<br>Photosensitiza<br>tion/<br>Completed<br>Challenge | Population II – Local Tolerability / Completed Induction but not Challenge | Population<br>III – AE<br>Safety/All<br>Subjects who<br>Received<br>Treatment |
| XX | XXXX-XX-XX | XXXX-XX-XX | XXXX-XX-XX (X) | | COMPLETED | XX | Y | Y | Y |
| XX | XXXX-XX-XX | XXXX-XX-XX | XXXX-XX-XX (X) | | COMPLETED | XX | Y | Y | Y |
| XX | XXXX-XX-XX | XXXX-XX-XX | XXXX-XX-XX (X) | XXXX-XX-XX (X) | SUBJECT IS LOST TO<br>FOLLOW-UP | XX | Y | Y | Y |
| XX | XXXX-XX-XX | XXXX-XX-XX | XXXX-XX-XX (X) | XXXX-XX-XX (X) | COMPLETED | XX | Y | Y | Y |
| XX | XXXX-XX-XX | XXXX-XX-XX | XXXX-XX-XX (X) | · , | INVESTIGATOR'S<br>JUDGEMENT | XX | Y | Y | Y |

<sup>[1]</sup> Study day is relative to Day 1.

Population I: Photosensitization potential for each test product site will be assessed only among subjects completing the Induction and Challenge Phases for that product.

Population II: Photoirritation potential for each test product will be assessed only among subjects completing the Induction Phase.

<sup>[2]</sup> Number of Days in Study is calculated as Date of Last Visit minus Date of Day 1 plus 1.

Population III: This population will include all subjects who received the study products.


# Listing 16.2.2: Protocol Deviations All Randomized Subjects

| Subject Number | Protocol Deviation Description | Туре | Action Taken |
|---|---|---|---|
| XX | xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx | xxxxxxxxx | xxxxx |
| XX | xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx | xxxxxxxxx | xxxxx |
| XX | xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx | xxxxxxxxx | XXXXX |

MC2 Therapeutics


Listing 16.2.4.1: Demographics and Baseline Characteristics
All Randomized Subjects

| Subject<br>Number | Date of Birth | Age<br>(Years) [1] | Gender | Race | Ethnicity | Fitzpatrick Skin Type [2] |
|---|---|---|---|---|---|---|
| XX | xxxx-xx-xx | xx | xxxxxx | xxxxxxxxxx | xxxxxxxxxxxxxxxxx | I |
| XX<br>XX | XXXX-XX-XX<br>XXXX-XX-XX | XX<br>XX | XXXXXX<br>XXXXXX | xxxxxx<br>Multiple: xxxxxxxxxxxxx | xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx | III<br>II |
| xx | xxxx-xx-xx | XX | XXXXXX | XXXXXX | xxxxxxxxxxxxxxxxxx | I |

Generated on XX/XX/XX:XXXX by XXXXXXX / Uses: XXXX, XXXX

Page X of Y

<sup>[1]</sup> Age is relative to Day 1.

<sup>[2]</sup> I = Always burns easily, never tans; II = Always burns easily, tans minimally; III = Burns moderately, tans gradually


Listing 16.2.4.2: Medical History All Randomized Subjects

| Subject<br>Number | Diagnosis and/or Procedure | Onset Date | Resolution Date |
|---|---|---|---|
| xx | xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx | XXXX<br>XXXX-XX-XX | XXXX-XX-XX<br>Ongoing |
| XX | xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx | XXXX-XX-XX | XXXX-XX-XX |
| XX | xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx | XXXX-XX | Ongoing |


# Listing 16.2.4.3: Prior and Concomitant Medications All Randomized Subjects

| Subject<br>Number | WHO Preferred Term (Verbatim Term)/ ATC Classification | Indication<br>Dose / Unit / Route / Frequency | Start Date (Day) – Stop Date (Day) |
|---|---|---|---|
| | XXXXXXXX (XXXXXXXXXXXXXXXXXXXXXXXXXXXX | XXXXXXXXXXXXX | |
| XX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XXXXX / XX / XXXX/ XXXX | XXXX-XX-XX(XX) - XXXX-XX-XX(XX) |
| | XXXXXXXX (XXXXXXXXXXXXXXXXXXXXXXXXXXXX | XXXXXXXXXXXXX | |
| | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XXXXX / XX / XXXX/ XXXX | XXXX – Ongoing |
| | XXXXXXXX (XXXXXXXXXXXXXXXXXXXXXXXXXXXX | xxxxxxxxxxxx | |
| XX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XXXXX / XX / XXXX/ XXXX | XXXX – XXXX-XX-XX (XX) |

Note: Study day is calculated relative to Baseline (Day 1).

MC2 Therapeutics Protocol No. MC2-01-C10

Page X of Y

# Listing 16.2.5: MED Determination All Randomized Subjects

| | | | | | | Subsite | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Subject<br>Number | Date-Time of<br>Irradiation | Time Point Post-<br>Irradiation Date-Time of Reading | Date-Time of Reading | | 1 | 2 | 3 | 4 | 5 | 6 | MED |
| XX | xxxx-xx-xxTxx:xx | | | UVB/UVA Intensity (μW/cm²) | xx | XX | XX | XX | XX | XX | |
| | | | | Exposure (seconds) | XX | XX | XX | XX | XX | XX | |
| | | Immediate | xxxx-xx-xxTxx:xx | Reading | XX | XX | XX | XX | XX | XX | |
| | | 16 – 24 Hours | xxxx-xx-xxTxx:xx | Reading | XX | XX | XX | XX | XX | XX | X.XX |
| xx | xxxx-xx-xxTxx:xx | | | UVB/UVA Intensity (μW/cm²) | XX | xx | XX | XX | xx | XX | |
| | | | | Exposure (seconds) | XX | XX | XX | XX | XX | XX | |
| | | Immediate | xxxx-xx-xxTxx:xx | Reading | XX | XX | XX | XX | XX | XX | |
| | | 16 – 24 Hours | xxxx-xx-xxTxx:xx | Reading | XX | XX | XX | XX | XX | XX | X.XX |


## Listing 16.2.6.1: Assessment of Dermal Responses During Induction Population II

| | Date-Time UVB/UV | | MC2-01 cream | | MC2-01 vehicle | | Untreated | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| Subject | of | A | 2xMED | Time | Date-Time of | | Non- | | Non- | |
| Number | Application | $(\mu W/cm^2)$ | (seconds) | Point | Reading | Irradiated | Irradiated | Irradiated | Irradiated | Irradiated |
| | | | | | | ER/ED (Sum) | ER/ED (Sum) | ER/ED (Sum) | ER/ED (Sum) | ER/ED (Sum) |
| XX | xxxx-xx-<br>xxTxx:xx | X.XX | X.XX | Day 2 | xxxx-xx-xxTxx:xx | x/y (Sum) | x/y (Sum) | x/y (Sum) | x/y (Sum) | x/y (Sum) |
| | | | | Day 4 | xxxx-xx-xxTxx:xx | x/y (Sum) | x/y (Sum) | x/y (Sum) | x/y (Sum) | x/y (Sum) |
| | | | | Day 5 | xxxx-xx-xxTxx:xx | x/y (Sum) | x/y (Sum) | x/y (Sum) | x/y (Sum) | x/y (Sum) |
| | | | | Day 8 | xxxx-xx-xxTxx:xx | x/y (Sum) | x/y (Sum) | x/y (Sum) | x/y (Sum) | x/y (Sum) |
| | | | | Day 9 | xxxx-xx-xxTxx;xx | x/y (Sum) | x/y (Sum) | x/y (Sum) | x/y (Sum) | x/y (Sum) |
| | | | | etc. | | | | | | |
| | | | Mean Pate | ch Response | e Score | XX | XX | XX | XX | XX |
| | | | | etc | | | | | | |

#### **Scores:**

 $Erythema;\ 0 = No\ reaction;\ 1 = Mild,\ but\ definite\ erythema;\ 2 = Moderate\ erythema;\ 3 = Marked/severe\ erythema;$ 

Edema: 0 = No reaction; 1 = Mild, but definite edema; 2 = Definite edema with erosion/vesiculation

#### **Notations:**

Hr = hyperpigmentation; Ho = hypopigmentation; V = vesiculation; p= Papular response; pv= Papulovesicular response; D= Damage to epidermis; oozing, crusting, and/or superficial erosions; I=Itching; S= Spreading of reaction beyond patch study site (i.e., reaction where material did not contact skin); f= Follicular irritation with or without pustule formation (folliculitis).; X=Subject absent; PD=Patch dislodged; NP = Not Patched; 0=No Reaction

 $[Programming\ Note:\ Present\ Notation\ if\ applicable\ after\ erythema\ and\ edema\ scores,\ in\ the\ format:\ ER/ED/NOTATION\ (Sum).]$ 

Generated on  $\ XX/XX/XX:XXXX\$  by  $\ XXXXXXX\$  / Uses:  $\ XXXX,\ XXXX$ 

[A similar listing will be produced for Residual Dermal Responses at Relocated Treatment Sites if Necessary (Listing 16.2.6.2)]

MC2 Therapeutics

Page X of Y

Listing 16.2.6.3: Assessment of Dermal Responses During Challenge All Randomized Subjects

| | | UVB | | 1/ MED | 6 | Time | | MC2-0 | 1 cream | MC2-0 | 1 vehicle | Untreated |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Subject<br>Number | Date-Time of<br>Application | /UVA<br>(μW/<br>cm²) | UVA<br>(mW/<br>cm²) | ½ MED<br>UVB/U<br>VA<br>(sec) | J/cm <sup>2</sup><br>UVA<br>(sec) | Point<br>Post-<br>Irradia<br>tion | Date-Time<br>of Reading | Irradiated | Non-<br>Irradiated | Irradiated | Non-<br>Irradiated | Irradiated |
| | | | | | | | | ER/ED (Sum) | ER/ED (Sum) | ER/ED (Sum) | ER/ED (Sum) | ER/ED (Sum) |
| XX | xxxx-xx-<br>xxTxx:xx | X.XX | XX.XX | XX.XX | XX.XX | 0 hrs<br>24 hrs | xxxx-xx-xx<br>Txx:xx<br>xxxx-xx-xx<br>Txx:xx | x/y (Sum)<br>x/y (Sum) | x/y (Sum) x/y (Sum) | x/y (Sum) x/y (Sum) | x/y (Sum) x/y (Sum) | x/y (Sum)<br>x/y (Sum) |
| | | | | | | 48 hrs<br>72 hrs | xxxx-xx-xx<br>Txx:xx<br>xxxx-xx-xx | x/y (Sum) | x/y (Sum) | x/y (Sum) | x/y (Sum) | x/y (Sum) |
| | | | | | Photos | sensitized ( | Txx:xx<br>Yes/No) [1] | x/y (Sum)<br>No | x/y (Sum)<br>No | x/y (Sum)<br>No | x/y (Sum)<br>No | x/y (Sum)<br>No |

[1] Sensitization classification made by the PI based on Challenge and Re-challenge

#### Scores:

Erythema: 0 = No reaction; 1 = Mild, but definite erythema; 2 = Moderate erythema; 3 = Marked/severe erythema;

Edema: 0 = No reaction; 1 = Mild, but definite edema; 2 = Definite edema with erosion/vesiculation

#### **Notations:**

Hr = hyperpigmentation; Ho = hypopigmentation; V = vesiculation; p= Papular response; pv= Papulovesicular response; D= Damage to epidermis; oozing, crusting, and/or superficial erosions; I=Itching; S= Spreading of reaction beyond patch study site (i.e., reaction where material did not contact skin); f= Follicular irritation with or without pustule formation (folliculitis).; X=Subject absent; PD=Patch dislodged; NP = Not Patched; 0=No Reaction

[Programming Note: Present Notation if applicable after erythema and edema scores, in the format: ER/ED/NOTATION (Sum).]

Generated on  $\ XX/XX/XX:XXXX\$  by  $\ XXXXXXX\$  / Uses:  $\ XXXX,\ XXXX$ 

[Note: A similar listing will be produced for any Rechallenge Phase assessments as needed.]

**MC2** Therapeutics


Page X of Y

# Listing 16.2.7.1: Adverse Events Population III

| Subject<br>Number | MedDRA Term (Verbatim Term) /<br>MedDRA SOC Term | Treatment-emergent? / Date (Day) of Onset – Date of Resolution (Day) | Intensity /<br>Relationship /<br>Outcome | Action Taken with Study Drug / Action Taken to Treat the Event? / Serious Adverse Event (SAE)? |
|---|---|---|---|---|
| xx | xxxxxxxxx (xxxxxxxxxxxxxxxxxxxxxxxxxxx | Yes / xxxx-xx-xx (xx) - xxxx-xx-xx (xx) No / xxxx-xx-xx (xx) - Ongoing | Severe / Possibly Related / Recovering Mild / Not related / Recovered | Dose reduced / Yes / Yes Dose not changed / No / No |
| XX | xxxxxxxxx (xxxxxxxxxxxxxxxxxxxxxxxxxxx | Yes /<br>xxxx-xx-xx (xx) – xxxx-xx-xx (xx) | Moderate /<br>Probably Related /<br>Recovered | Dose not changed /<br>No /<br>No |

Note: A treatment-emergent AE is an AE with an onset date on or after the first study product administration date. Study day is relative to Day 1.


# Listing 16.2.7.2: Serious Adverse Events and Deaths All Randomized Subjects

| Subject Number | MedDRA Term (Verbatim Term) / MedDRA SOC Term | Treatment-emergent? / Date (Day) of Onset – Date of Resolution (Day) | Intensity /<br>Relationship /<br>Outcome | Action Taken with Study Drug / Action Taken to Treat the Event?/ Which Serious Criteria Met? |
|---|---|---|---|---|
| xx | xxxxxxxxx (xxxxxxxxxxxxxxxxxxxxxxxxxxx | Yes / xxxx-xx-xx (xx) - xxxx-xx-xx (xx) No / xxxx-xx-xx (xx) - Ongoing | Severe /<br>Possibly Related /<br>Recovering<br>Severe /<br>Not related /<br>Recovering | Dose reduced / Yes / Life Threatening Drug withdrawn / Yes / Hospitalization |
| XX | xxxxxxxxx (xxxxxxxxxxxxxxxxxxxxxxxxxxx | Yes / xxxx-xx-xx (xx) – xxxx-xx-xx (xx) | Moderate /<br>Probably related /<br>Recovered | Drug withdrawn /<br>Yes /<br>Other Medically Serious Event |

Note: A treatment-emergent AE is an AE with an onset date on or after the first study product administration date. Study day is relative to Day 1.


# Listing 16.2.8: Urine Pregnancy Test Results All Randomized Subjects

| | _ | Urine Pregnancy Test | | | |
|---|---|---|---|---|---|
| Subject | | Day | y 1 | End of Study | |
| Number | Childbearing Potential | Date | Result | Date | Result |
| XX | xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx | xxxx-xx-xx | Negative | xxxx-xx-xx | Negative |
| XX | Postmenopausal | | N/A | | N/A |
| XX | N/A (Male Subject) | | N/A | | N/A |

Note: NA for males/females of non-childbearing potential.

MC2 Therapeutics Protocol No. MC2-01-C10

Page X of Y

Listing 16.2.9: Comments All Randomized Subjects

| Subject<br>Number | Reference | Comment |
|---|---|---|
| XX | GENERAL COMMENTS<br>END OF STUDY | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX |
| xx | GENERAL COMMENTS | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX |